CLINICAL TRIAL: NCT03318900
Title: Phase I/Ib Study of Adoptive Cellular Therapy Using Autologous IL-21-Primed CD8+ Tumor Antigen-Specific T Cells in Combination With Utomilumab (PF-05082566) in Patients With Platinum Resistant Ovarian Cancer
Brief Title: T-Cell Infusion, Aldesleukin, and Utomilumab in Treating Patients With Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0400; NCI-2018-01034 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0400 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-10-16; First posted 2017-10-24 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: COL6A3 Positive; HLA-A*0201 Positive Cells Present; PRAME Positive; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — aldesleukin; CD8 antigen, alpha chain; CD8 Antigens; Cyclophosphamide; Leukapheresis; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (T-cell infusion, aldesleukin, utomilumab) (Experimental): Patients undergo leukapheresis. Patients then receive cyclophosphamide IV on day -2, CD8-positive T-lymphocyte via infusion on day 0, and aldesleukin SC every 12 hours for 14 days. Beginning 24 hours after CD8-positive T-lymphocyte, patients also receive utomilumab IV over 90 minutes on days 1, 29, 57, 85, 113, and 141 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Drug: CD8-Positive T-Lymphocyte; Drug: Cyclophosphamide; Procedure: Leukapheresis; Biological: Utomilumab

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: CD8-Positive T-Lymphocyte — Given IV
  Other Names: CD8 Cell; CD8 Lymphocyte; CD8 Lymphocytes; CD8+ T Cell; CD8+ T Lymphocyte; CD8+ T Lymphocytes; CD8+ T-Lymphocyte; CD8-Positive Lymphocyte; CD8-Positive Lymphocytes; CD8-Positive T-Lymphocytes; T8 Cell; T8 Cells; T8 Lymphocyte; T8 Lymphocytes
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Biological: Utomilumab — Given IV
  Other Names: PF 05082566; PF 5082566; PF-05082566; PF-2566

SUMMARY:
This phase I/Ib trial studies the side effects and best dose of utomilumab and how well it works with CD8-positive T-lymphocyte (T-cell infusion) and aldesleukin in treating patients with ovarian cancer that has come back. Aldesleukin may stimulate white blood cells to kill ovarian cancer cells. Giving white blood cells (T-cells) that have been activated by a vaccine with aldesleukin may kill more tumor cells. Immunotherapy with utomilumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving T-cell infusion with aldesleukin and utomilumab may work better in treating patients with ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and toxicity of adoptively transferred central memory-type CTL targeting ovarian cancer antigens administered alone, and in combination with, utomilumab, an agonistic anti-CD137 antibody, in patients with platinum-resistant ovarian cancer.

II. Evaluate the functional and numeric in vivo persistence of adoptively transferred central memory-type CTL with and without utomilumab.

SECONDARY OBJECTIVES:

I. Evaluate the anti tumor effect of adoptively transferred central memory-type CTL targeting ovarian cancer antigens as measured by best overall response rate (BORR) and progression free survival (PFS).

OUTLINE: This is a dose escalation study of utomilumab.

Patients undergo leukapheresis. Patients then receive cyclophosphamide intravenously (IV) on day -2, CD8-positive T-lymphocyte via infusion on day 0, and aldesleukin subcutaneously (SC) every 12 hours for 14 days. Beginning 24 hours after CD8-positive T-lymphocyte, patients also receive utomilumab IV over 90 minutes on days 1, 29, 57, 85, 113, and 141 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 3, 7, 14, 22, 28, 35, 43, 49, 56, 64, 70, 77, 84, 112, and 140.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic documentation (must be performed or reviewed at MD Anderson) of recurrent high grade epithelial ovarian cancer.
* At least one prior line of platinum-based chemotherapy (subjects are eligible for enrollment and leukapheresis while still platinum-sensitive, however, they must have developed platinum resistant disease for treatment (turnstile 2).
* Tumor expressing PRAME and/or COL6A3.
* Expression of HLA-A*0201.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Expected survival of greater than 16 weeks.
* Willing and able to give informed consent.
* Hemoglobin >= 9.0 g/dL.
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (>=1000 per mm^3).
* Platelet count >= 75 x 10^9/L (>=100,000 per mm^3).
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN) unless diagnosed with Gilbert's syndrome.
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN unless liver metastases are present, in which case it must be =< 5x ULN.
* Serum creatinine clearance (CL) >40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance.
* Subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 50 years old and no menses for >=1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized. Suggested precautions should be used to minimize the risk or pregnancy for at least 1 month before start of therapy, and while women are on study for up to 3 months after T cell infusion, and at least 8 weeks after the study drug is stopped.
* {Turnstile 2} Subjects must have platinum resistant disease (progression on a platinum-containing regimen or recurrence within 180 days of last dose of platinum-containing chemotherapy). Subjects that are not platinum resistant but are deemed not to be candidates for platinum-based chemotherapy due to prior significant allergic reaction may participate with principal investigator (PI) approval.
* {Turnstile 2} Bi-dimensionally measurable disease by radiographic imaging (magnetic resonance imaging [MRI] or computed tomography [CT] scan).
* {Turnstile 2} At least 4 weeks must have elapsed since the last chemotherapy, immunotherapy, radiotherapy or major surgery. At least 6 weeks for bevacizumab.
* {Turnstile 2} Toxicity related to prior therapy must either have returned to =< grade 1, baseline, or been deemed irreversible.

Exclusion Criteria:

* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam. Patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in one second (FEV1) < 60% of normal or carbon monoxide diffusing capacity (DLco) (corrected [corr] for hemoglobin [Hgb]) < 55% will be excluded.
* Significant cardiovascular abnormalities including any one of the following: Congestive heart failure, Clinically significant hypotension, symptoms of coronary artery disease, presence of cardiac arrhythmias on electrocardiography (EKG) requiring drug therapy; or patients with a history of cardiovascular disease. (Patients with the above will undergo a cardiac evaluation which can include a stress test and/or echocardiography. Results of this evaluation will be considered before excluding patients on the basis of cardiovascular abnormalities). Subjects with evidence of stress-induced cardiac ischemia or ejection fraction less than 55% will be excluded.
* History of central nervous system (CNS) metastasis.
* Autoimmune disease: patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of autoimmune disease (e.g. systemic lupus erythematosus, vasculitis, infiltrating lung disease) whose possible progression during treatment would be considered by the Investigator to be unacceptable.
* {Turnstile 2} Participation in another clinical study with an investigational product administered during the last 28 days.
* {Turnstile 2} Receipt of the last dose of previous chemotherapy, hormonal, or biologic treatment for ovarian, fallopian tube, or primary peritoneal cancer in the last 28 days (in the last 6 weeks for bevacizumab).
* {Turnstile 2} Current or prior use of immunosuppressive medication within 28 days before enrollment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* {Turnstile 2} Any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1.
* History of allogeneic organ transplant.
* Unresolved partial or complete small or large bowel obstruction.
* {Turnstile 2} Receipt of live attenuated vaccination within 30 days prior to enrollment or within 30 days of planned lymphodepletion.
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events.
* Active viral hepatitis.
* Confirmed human immunodeficiency virus (HIV) infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir A Jazaeri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 07/16/2018 and the first participant was enrolled on 09/04/2018. The study was completd on 09/04/2020 when the last particiapnt treated was taken off study and the study was terminated on 12/20/2023. All screening and recruitment was done in a medical clinic setting.
Groups:
- Dose Level 1: Cyclophosphamide (300 mg/m2) IV 2 days prior to infusion of T-Cells IV on Day 0 followed by IL-2 SC injections every 12 hours for 14 days
- Dose Level 2: Cyclophosphamide (300 mg/m2) IV 2 days prior to infusion of T Cells IV on Day 0 followed by IL-2 SC injections every 12 hours for 14 days; low-dose anti-CD137 IV beginning on Day 1 and then every 4 weeks x6 doses
- Dose Level 3: Cyclophosphamide (300 mg/m2) IV 2 days prior to infusion of T Cells IV on Day 0 followed by IL-2 SC injections every 12 hours for 14 days; high-dose anti-CD137 IV beginning on Day 1 and then every 4 weeks x6 doses
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Started | 3 | 2 | 0
Completed | 3 | 2 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to lack of funding, dose level 3 did not recruit any participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Total
Number analyzed (Participants) | 3 | 2 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 0 | 5
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Assess Safety and Toxicity of Adoptively Transferred Central Memory-type CTL Targeting Ovarian Cancer Antigens Administered Alone, and in Combination With, Utomilumab, an Agonistic Anti-CD137 Antibody, in Patients With Platinum Resistant Ovarian Cancer
Description: Due to lack of funding, the study was not able to accrue a sample size large enough to address the primary and secondary objectives
Time Frame: will continue to be monitored on study with visits every 8 weeks or as often as clinically indicated unless the disease gets worse, participants starts another therapy, or the participants are taken off study
Population: Data were not collected due to lack of funding; the study was not able to accrue a sample size large enough to address the primary and secondary objectives
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Evaluate the Anti Tumor Effect of Adoptively Transferred Central Memory-type CTL Targeting Ovarian Cancer Antigens as Measured by Best Overall Response Rate (BORR) and Progression Free Survival (PFS).
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 18 months
Description: CTCAE V5.0
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=2) | Dose Level 3 (N=0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=2) | Dose Level 3 (N=0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03318900/Prot_SAP_001.pdf